CLINICAL TRIAL: NCT02059811
Title: Efficacy and Safety of the Dietary Approaches to Stop Hypertension (DASH) Diet in Adults With Moderate Chronic Kidney Disease: Pilot Study
Brief Title: Efficacy and Safety of the DASH Diet in Adults With Moderate Chronic Kidney Disease: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00048112
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Hypertension; Chronic Kidney Disease
Keywords: Kidney Diseases; Renal Insufficiency, Chronic; Diet; DASH diet; Hypertension; Vascular diseases; Cardiovascular Diseases; Blood pressure
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic; Kidney Diseases; Vascular Diseases; Cardiovascular Diseases | interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DASH Diet (Experimental): All participants will be provided a control diet for a 7-day run-in period followed by the DASH dietary intervention for a 14-day intervention period. Participants will consume the largest meal of the day in a supervised setting at the study center and all other meals and snacks will be provided in "to-go" packages. Weight will be held constant by measuring participant weight daily and adjusting caloric content of meals. Adherence will be monitor by review of daily food diaries.
  Interventions: Other: DASH Diet; Other: Control Diet

INTERVENTIONS:
Other: DASH Diet — The DASH diet is a nutritional intervention that is low in cholesterol and saturated fat and emphasizes high intake of the following: fruits, vegetables, low-fat dairy products, whole grains, fiber, and protein derived mostly from plant sources.
Other: Control Diet — The control diet, which is a diet typical of most Americans, is relatively high in total and saturated fat and cholesterol, and low in servings of fruits, vegetables and low fat dairy products.

SUMMARY:
More than two-thirds of US adults with chronic kidney disease (CKD) have uncontrolled hypertension. Both hypertension and CKD are major independent risk factors for cardiovascular disease, which is the leading cause of death in the US. Fortunately, lowering blood pressure to recommended treatment targets not only slows the progression of CKD, but also improves cardiovascular outcomes. Controlling hypertension in this patient population, however, can be quite challenging. A lifestyle modification that effectively reduces blood pressure in both pre-hypertensive and hypertensive adults is the Dietary Approaches to Stop Hypertension (DASH) diet.

The purpose of this pilot study is to (1) determine the extent to which the DASH diet lowers blood pressure in hypertensive adults with moderate chronic kidney disease (CKD) (estimated glomerular filtration rate [eGFR] 30-59 ml/min/1.73m2) and (2) establish that the DASH diet can be safely consumed by this patient population.

DETAILED DESCRIPTION:
During a 7-day run-in phase, participants will first consume a control diet similar in nutrient composition to the control diet of previous DASH studies. The control diet, which is a diet typical of most Americans, is reduced in servings of fruits, vegetables, low fat dairy products and relatively high in total and saturated fat. Immediately following the run-in phase, participants will receive the DASH diet during a 14-day intervention phase. Both diets will have the same sodium content and caloric intake will be adjusted for each participant to keep weight stable. All study meals and snacks will be provided.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* eGFR 30-59 ml/min/1.73m2
* SBP ≥ 130 mmHg or DBP ≥ 80 mmHg
* willing to eat one meal on-site 5 days/week

Exclusion Criteria:

* baseline potassium >4.6 mEq/L while not taking potassium supplements (if potassium is ≥ 5.0 while taking potassium supplements, a potassium of 4.6 or less must be demonstrated off supplements
* evidence of hyperkalemia (>5.1 mEq/L) within last 6 months
* ≥ 0.5 mg/dl increase in serum creatinine in past 6 months
* albumin-to-creatinine ratio > 200 mg/mmol
* insulin requiring or poorly controlled diabetes mellitus
* cardiovascular event within previous 6 months
* change in anti-hypertensive medications in last 2 weeks, or anticipated medication change during study period
* unwillingness to eat only study food for 21 day study period
* unwillingness or inability to discontinue vitamin and mineral supplements or antacids containing potassium, magnesium or calcium
* use of aldosterone antagonist
* use of oral corticosteroids
* alcohol intake >14 drinks/week
* unstable doses of psychotropics or phenothiazine
* weight reducing medications
* use of medications for erectile dysfunction during study period
* pregnant, breast feeding, or planning pregnancy during study period
* chronic disease that may interfere with participation
* history of organ transplant
* any serious illness that would interfere with participation or make DASH diet unsafe
* planning to leave the area during the study period
* significant food allergies, preferences, or dietary requirements that would interfere with diet adherence
* investigator discretion for safety or compliance reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in office systolic blood pressure | 2 weeks post DASH diet intervention
  A comparison of pre-intervention and post-intervention systolic blood pressure will be completed.

SECONDARY OUTCOMES:
Change in serum potassium | 2 weeks post DASH diet intervention
  A comparison of pre-intervention and post-intervention serum potassium will be completed.

OTHER OUTCOMES:
Change in blood pressure | 2 weeks post DASH diet intervention
  A comparison of pre-intervention and post-intervention office diastolic blood pressure and 24 hour ambulatory systolic and diastolic blood pressure will be completed.
Change in markers of kidney function | 2 weeks post DASH diet intervention
  A comparison of pre-intervention and post-intervention markers of kidney function (creatinine, eGFR, and urine albumin-to-creatinine ratio) will be completed.
Change in markers of mineral metabolism | 2 weeks post DASH diet intervention
  A comparison of pre-intervention and post-intervention markers of mineral metabolism (calcium, phosphorus, intact parathyroid hormone, and 25-hydroxyvitamin D) will be completed.
Change in serum electrolytes | 2 weeks post DASH diet intervention
  A comparison of pre-intervention and post-intervention electrolytes (bicarbonate, urea nitrogen) will be completed.
Change in fasting glucose | 2 weeks post DASH diet intervention
  A comparison of pre-intervention and post-intervention fasting glucose will be completed.
Change in 24 hour urinary excretion | 2 weeks post DASH diet intervention
  A comparison of pre-intervention and post-intervention urinary excretion of sodium, potassium, urea nitrogen, calcium, phosphorus, magnesium, creatinine, and albumin will be completed.

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Tyson, MD, Principal Investigator — Duke University
Locations (1):
- Stedman Nutrition and Metabolism Center, Center for Living, Durham, North Carolina, United States